CLINICAL TRIAL: NCT02330874
Title: Assessment of the Risk of Unplanned Readmission to the Intensive Care Unit Using the Safe Discharge From ICU (SD-ICU) Score: A Validation Study.
Brief Title: Validation of the SD-ICU. A Risk Assessment Tool of Unplanned ICU Readmission
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, PhD, Hospital Sao Domingos
Other Study IDs: 003/2014
Record Dates: First submitted 2014-12-28; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Critical Illness
Keywords: Risk; score; readmission; ICU
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In a recent study, which included 845 patients that at the time of ICU discharge had at least one risk factor for readmission, the investigators' group developed a new readmission risk score in the ICU, Safe Discharge from ICU (SD-ICU), using parameters easily and routinely measured in ICU: the Charlson comorbidity (ICC), the TISS-28 (Therapeutic Intervention Scoring System - 28), the length of stay in ICU and age. Through ROC curve analysis, the investigators found that patients with a score above 14.5 had a high probability of readmission.

The objective of this study is to validate the Safe Discharge from ICU (SD-ICU) score as a tool to predict unplanned readmissions to the intensive care unit.

All adult patients discharged from a 37 bed general ICU from April 2014 to March 2015 will be included in the study. The SD-ICU score is routinely calculated at the time of discharge from the ICU. Patients will be divided into two groups: those with SD-ICU score> 14.5 (group 1) and those with a score equal to or less than 14.5 (group 2). The two groups will be compared with respect to the frequency of unplanned readmissions. Stepwise, multivariate logistic regression will be used to investigate the association between the risk factors for readmission used in SD-ICU score and ICU readmission as outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients discharged from a general ICU

Exclusion Criteria:

* Patients under 18 years old
* Those that were not candidates for ICU readmission (interhospital and home care transfer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients discharged alive from a general ICU
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Readmission to the ICU | After ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, PhD, Principal Investigator — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil